CLINICAL TRIAL: NCT00083603
Title: A Phase I Trial to Evaluate the Safety and Immunogenicity of rMVA-HIV (rMVA-HIV Env/Gag + rMVA-HIV Tat/Rev/Nef-RT) and rFPV-HIV (rFPV-HIV Env/Gag + rFPV-HIV Tat/Rev/Nef-RT) Vaccines, Alone or in Combination, in Healthy, Vaccinia Naive HIV-1 Negative Participants
Brief Title: Safety of and Immune Response to Two HIV Vaccine Formulations (rMVA-HIV and rFPV-HIV) Alone or in Combination in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 055; 10056 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2004-05-26; First posted 2004-05-27 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine; Vaccinia vector; Pox vector
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (16):
- 1 (Experimental): rFPV-HIV vaccine administered as two separate 1-mL intramuscular injections, with rFPV-HIV env/gag into the left deltoid, rFPV-HIV tat/rev/nef-RT into the right deltoid at Days 0, 28, 84, 140, and 196
  Interventions: Biological: rFPV-HIV (rFPV-HIV env/gag + rFPV-HIV tat/rev/nef-RT)
- 2 (Placebo Comparator): Empty TBC-FPV vector administered as two separate 1-mL intramuscular injections, one into each deltoid at Days 0, 28, 84, 140, and 196
  Interventions: Biological: Empty TBC-FPV
- 3 (Experimental): rMVA-HIV env/gag and rMVA-HIV tat/rev/nef-RT administered as two separate 1-mL intramuscular injections, with rMVA-HIV env/gag into the left deltoid, rMVA-HIV tat/rev/nef-RT into the right deltoid at Days 0, 28; rFPV-HIV env/gag and rFPV-HIV tat/rev/nef-RT administered as two separate 1-mL intramuscular injections, with rFPV-HIV env/gag into the left deltoid, rFPV-HIV tat/rev/nef-RT into the right deltoid at Days 84, 140, and 196
  Interventions: Biological: rMVA-HIV (rMVA-HIV env/gag + rMVA-HIV tat/rev/nef-RT); Biological: rFPV-HIV (rFPV-HIV env/gag + rFPV-HIV tat/rev/nef-RT)
- 4 (Placebo Comparator): Empty TBC-MVA vector administered in each deltoid on Days 0, 28; empty TBC-FPV vector administered in each deltoid on Days 84, 140, and 196
  Interventions: Biological: Empty TBC-FPV; Biological: TBC-MVA and TBC-FPV
- 5 (Experimental): rMVA-HIV env/gag and rMVA-HIV tat/rev/nef-RT administered as two separate 1-mL intramuscular injections, with rMVA-HIV env/gag into the left deltoid, rMVA-HIV tat/rev/nef-RT into the right deltoid at Days 0, 28; rFPV-HIV env/gag and rFPV-HIV tat/rev/nef-RT administered as two separate 1-mL intramuscular injections, with rFPV-HIV env/gag into the left deltoid, rFPV-HIV tat/rev/nef-RT into the right deltoid at Days 84, 140, and 196
  Interventions: Biological: rFPV-HIV (rFPV-HIV env/gag + rFPV-HIV tat/rev/nef-RT); Biological: rMVA-HIV (rMVA-HIV env/gag + rMVA-HIV tat/rev/nef-RT)
- 6 (Placebo Comparator): Empty TBC-MVA vector administered in each deltoid Days 0, 28; empty TBC-FPV vector administered in each deltoid Days 84, 140, and 196
  Interventions: Biological: Empty TBC-FPV; Biological: TBC-MVA and TBC-FPV
- 7 (Experimental): rMVA-HIV env/gag and rMVA-HIV tat/rev/nef-RT administered as two separate 1-mL intramuscular injections, with rMVA-HIV env/gag into the left deltoid, rMVA-HIV tat/rev/nef-RT into the right deltoid at Days 0, 28; rFPV-HIV env/gag and rFPV-HIV tat/rev/nef-RT administered as two separate 1-mL intramuscular injections, with rFPV-HIV env/gag into the left deltoid, rFPV-HIV tat/rev/nef-RT into the right deltoid at Days 84, 140, and 196
  Interventions: Biological: rFPV-HIV (rFPV-HIV env/gag + rFPV-HIV tat/rev/nef-RT); Biological: rMVA-HIV (rMVA-HIV env/gag + rMVA-HIV tat/rev/nef-RT)
- 8 (Placebo Comparator): Empty TBC-MVA vector administered in each deltoid Days 0, 28; empty TBC-FPV vector administered in each deltoid Days 84, 140, and 196
  Interventions: Biological: Empty TBC-FPV; Biological: TBC-MVA and TBC-FPV
- 9 (Experimental): rMVA-HIV env/gag and rMVA-HIV tat/rev/nef-RT administered as two separate 1-mL intramuscular injections, with rMVA-HIV env/gag into the left deltoid, rMVA-HIV tat/rev/nef-RT into the right deltoid at Days 0, 28, 84, 140, 196
  Interventions: Biological: rMVA-HIV (rMVA-HIV env/gag + rMVA-HIV tat/rev/nef-RT)
- 10 (Placebo Comparator): Empty TBC-MVA vector administered in each deltoid Days 0, 28, 84, 140, 196
  Interventions: Biological: TBC-MVA and TBC-FPV
- 11 (Experimental): rFPV-HIV vaccine administered as two separate 1-mL intramuscular injections, with rFPV-HIV env/gag into the left deltoid, rFPV-HIV tat/rev/nef-RT into the right deltoid at Days 0, 28, 84, 140, and 196
  Interventions: Biological: rFPV-HIV (rFPV-HIV env/gag + rFPV-HIV tat/rev/nef-RT)
- 12 (Placebo Comparator): Empty TBC-FPV vector administered as two separate 1-mL intramuscular injections, one into each deltoid at Days 0, 28, 84, 140, and 196
  Interventions: Biological: Empty TBC-FPV
- 13 (Experimental): rMVA-HIV env/gag and rMVA-HIV tat/rev/nef-RT administered as two separate 1-mL intramuscular injections, with rMVA-HIV env/gag into the left deltoid, rMVA-HIV tat/rev/nef-RT into the right deltoid at Days 0, 28; rFPV-HIV env/gag and rFPV-HIV tat/rev/nef-RT administered as two separate 1-mL intramuscular injections, with rFPV-HIV env/gag into the left deltoid, rFPV-HIV tat/rev/nef-RT into the right deltoid at Days 84, 140, and 196
  Interventions: Biological: rFPV-HIV (rFPV-HIV env/gag + rFPV-HIV tat/rev/nef-RT); Biological: rMVA-HIV (rMVA-HIV env/gag + rMVA-HIV tat/rev/nef-RT)
- 14 (Placebo Comparator): Empty TBC-MVA vector administered in each deltoid Days 0, 28; empty TBC-FPV vector administered in each deltoid Days 84, 140, and 196
  Interventions: Biological: Empty TBC-FPV; Biological: TBC-MVA and TBC-FPV
- 15 (Experimental): rMVA-HIV env/gag and rMVA-HIV tat/rev/nef-RT administered as two separate 1-mL intramuscular injections, with rMVA-HIV env/gag into the left deltoid, rMVA-HIV tat/rev/nef-RT into the right deltoid at Days 0, 28, 84, 140, 196
  Interventions: Biological: rMVA-HIV (rMVA-HIV env/gag + rMVA-HIV tat/rev/nef-RT)
- 16 (Placebo Comparator): Empty TBC-MVA vector administered in each deltoid Days 0, 28, 84, 140, 196
  Interventions: Biological: TBC-MVA and TBC-FPV

INTERVENTIONS:
Biological: rMVA-HIV (rMVA-HIV env/gag + rMVA-HIV tat/rev/nef-RT) — rMVA 10^7 pfu /2mL administered in each deltoid
  Arms: 3
Biological: rFPV-HIV (rFPV-HIV env/gag + rFPV-HIV tat/rev/nef-RT) — Vaccines administered as two separate 1-mL intramuscular injections, with rFPV-HIV env/gag into the left deltoid, rFPV-HIV tat/rev/nef-RT into the right deltoid
  Arms: 1; 11; 13; 3; 5; 7
Biological: Empty TBC-FPV — Empty FPV 10^9 pfu/2mL administered as two separate 1 mL intramuscular injections, one into each deltoid.
  Arms: 12; 14; 2; 4; 6; 8
Biological: rMVA-HIV (rMVA-HIV env/gag + rMVA-HIV tat/rev/nef-RT) — rMVA 10^8 pfu /2mL administered in each deltoid
  Arms: 5
Biological: rMVA-HIV (rMVA-HIV env/gag + rMVA-HIV tat/rev/nef-RT) — rMVA 10^9 pfu /2mL administered in each deltoid
  Arms: 13; 15; 7; 9
Biological: TBC-MVA and TBC-FPV — Empty MVA 10^7 pfu/2mL administered into each deltoid
  Arms: 4
Biological: TBC-MVA and TBC-FPV — Empty MVA 10^8 pfu/2mL administered into each deltoid
  Arms: 6
Biological: TBC-MVA and TBC-FPV — Empty MVA 10^9 pfu/2mL administered into each deltoid
  Arms: 10; 14; 16; 8

SUMMARY:
The purpose of this study is to evaluate the safety of and immune response to two HIV vaccine formulations, rMVA-HIV and rFPV-HIV, alone and in combination, in HIV uninfected adults.

DETAILED DESCRIPTION:
Pox viruses are used for investigational vaccines in humans because they can accommodate large amounts of foreign DNA, can infect mammalian cells, and can access the cytotoxic T-cell responses believed to be important in the control of HIV infection and disease. Two pairs of matching recombinant HIV vaccines have been developed for use in this study. One pair uses a modified vaccinia Ankara (MVA) vector and the other pair uses a fowlpox vector (FPV). Each vaccine pair consists of one vaccine containing env/gag sequences and one vaccine containing modified tat/rev/nef-RT sequences. The HIV sequences are identical and are from a vertically transmitted pediatric primary isolate. The controls in this study are MVA vectors and FPVs without the HIV genes. The study will evaluate the safety and immunogenicity of the vaccine pairs.

There are two parts to this study. Participants in Part A will be randomly assigned to one of five different vaccination groups. Within each group, participants will be randomly assigned to receive either vaccine or control injections. Group 1 participants will receive the FPV vaccine pair or FPV control at each vaccine visit. Groups 2, 3, and 4 will receive one of three different doses of the MVA vaccine pair or MVA control at study entry and Month 1, then a fixed dose of the FPV vaccine pair or FPV control at Months 3, 5, and 7. Group 5 participants will receive the MVA vaccine pair or MVA control at maximum tolerated dose (MTD) at each vaccine visit. Groups 1 and 2 will enroll simultaneously; Groups 3, 4, and 5 will enroll as safety data from the previous groups become available.

In Part B, participants will be randomly assigned to receive study vaccine or control vaccine in one of three vaccination groups. Group 6 participants will receive the FPV vaccine pair or FPV control at each vaccine visit. Group 7 participants will receive the MVA vaccine pair or MVA control at study entry and Month 1, then a fixed dose of the FPV vaccine pair or FPV control at Months 3, 5, and 7. Group 8 participants will receive the MVA vaccine pair at MTD or MVA control at each vaccine visit. Enrollment into Groups 6, 7, and 8 will begin simultaneously after the completion of the safety data evaluation of Groups 1 and 2.

Study vaccinations will be given at study entry and at Months 1, 3, 5 and 7. Tests for cardiac injury will be performed at screening and at each 2-week follow-up visit after vaccination. Participants will have an electrocardiogram (ECG) at screening and 2 weeks after the first and last vaccinations. Study visits will occur at screening, study entry, and at 11 visits over 13 months. Study visits will consist of a physical exam, risk reduction/pregnancy prevention counseling, cardiac symptom assessment, and blood and urine collection. Women will have pregnancy tests at study entry and Months 1, 3, 5, 7, and 13.

ELIGIBILITY:
Note: As of 11/29/06, vaccinations in this trial have been discontinued.

Inclusion Criteria:

* HIV uninfected within 8 weeks prior to first vaccination
* Blood pressure 140/90 or less upon enrollment
* Good general health
* Willing to receive HIV test results
* Understand the vaccination procedure
* Negative for hepatitis B surface antigen
* Negative for anti-hepatitis C virus antibodies (anti-HCV) or negative for HCV PCR if anti-HCV is positive
* Willing to use acceptable forms of contraception
* Willing to be followed for the duration of the study
* Have access to a participating HIV vaccine trial site

Exclusion Criteria:

* HIV vaccines or placebos in prior HIV vaccine trial
* Previously received Avipox vaccine
* Previously received Vaccinia vaccine
* Immunosuppressive medications within 168 days prior to first vaccination
* Blood products within 120 days prior to first vaccination
* Immunoglobulin within 60 days prior to first vaccination
* Live attenuated vaccines within 30 days prior to first vaccination
* Investigational research agents within 30 days prior to first vaccination
* Medically indicated subunit or killed vaccines within 14 days prior to first study vaccine administration or allergy treatment with antigen injections within 30 days prior to first vaccination
* Current tuberculosis prophylaxis or therapy
* Hypersensitivity to egg products
* Past or present cardiac disease
* Two or more of the following cardiac risk factors: history of fasting LDL greater than 160 mg/dl; first degree relative who had heart condition, excluding hypertension; cigarette smoking
* ECG with clinically significant findings (e.g., conduction disturbance, repolarization abnormality, significant atrial or ventricular arrhythmia, frequent atrial or ventricular ectopy, ST elevation consistent with ischemia, evidence of past or evolving myocardial infarction)
* Serious adverse reaction to vaccines. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Unstable asthma
* Diabetes mellitus type 1 or 2
* Thyroid disease requiring treatment
* Serious angioedema within the last 3 years
* Bleeding disorder
* Malignancy unless it has been surgically removed and, in the opinion of the investigator, is not likely to recur during the study period
* Seizure disorder requiring medication within the past 3 years
* Absence of the spleen
* Mental illness that would interfere with the study
* Other conditions that, in the judgment of the investigator, would interfere with the study
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2004-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, as judged by local and systemic reactogenicity signs and symptoms, laboratory measures, and adverse events | After each injection and 12 months after the first injection
Immunogenicity, as judged by qualitative HIV-1-specific T-cell responses | At Days 98 and 210

CONTACTS AND LOCATIONS:
Overall Officials: Michael Keefer, MD, Study Chair — University of Rochester; Sharon Frey, MD, Study Chair — St. Louis University School of Medicine
Locations (6):
- United States (4):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - Saint Louis Univ. School of Medicine, HVTU, St Louis, Missouri
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - FHCRC/UW Vaccine CRS, Seattle, Washington
- Brazil (2):
  - Projeto Praça Onze/Hesfa Crs, Rio de Janeiro
  - Sao Paulo HVTU - CRT DST/AIDS CRS, São Paulo

REFERENCES:
- [Background] Amara RR, Villinger F, Altman JD, Lydy SL, O'Neil SP, Staprans SI, Montefiori DC, Xu Y, Herndon JG, Wyatt LS, Candido MA, Kozyr NL, Earl PL, Smith JM, Ma HL, Grimm BD, Hulsey ML, Miller J, McClure HM, McNicholl JM, Moss B, Robinson HL. Control of a mucosal challenge and prevention of AIDS by a multiprotein DNA/MVA vaccine. Science. 2001 Apr 6;292(5514):69-74. doi: 10.1126/science.1058915. PMID 11393868
- [Background] Blanchard TJ, Alcami A, Andrea P, Smith GL. Modified vaccinia virus Ankara undergoes limited replication in human cells and lacks several immunomodulatory proteins: implications for use as a human vaccine. J Gen Virol. 1998 May;79 ( Pt 5):1159-67. doi: 10.1099/0022-1317-79-5-1159. PMID 9603331
- [Background] Hanke T, McMichael AJ, Mwau M, Wee EG, Ceberej I, Patel S, Sutton J, Tomlinson M, Samuel RV. Development of a DNA-MVA/HIVA vaccine for Kenya. Vaccine. 2002 May 6;20(15):1995-8. doi: 10.1016/s0264-410x(02)00085-3. PMID 11983261
- [Background] Kent SJ, Zhao A, Best SJ, Chandler JD, Boyle DB, Ramshaw IA. Enhanced T-cell immunogenicity and protective efficacy of a human immunodeficiency virus type 1 vaccine regimen consisting of consecutive priming with DNA and boosting with recombinant fowlpox virus. J Virol. 1998 Dec;72(12):10180-8. doi: 10.1128/JVI.72.12.10180-10188.1998. PMID 9811759
- [Background] Stratov I, DeRose R, Purcell DF, Kent SJ. Vaccines and vaccine strategies against HIV. Curr Drug Targets. 2004 Jan;5(1):71-88. doi: 10.2174/1389450043490686. PMID 14738219
- [Result] Ramjee G, Kapiga S, Weiss S, Peterson L, Leburg C, Kelly C, Masse B; HPTN 055 Study Team. The value of site preparedness studies for future implementation of phase 2/IIb/III HIV prevention trials: experience from the HPTN 055 study. J Acquir Immune Defic Syndr. 2008 Jan 1;47(1):93-100. doi: 10.1097/QAI.0b013e31815c71f7. PMID 17984760
- [Derived] Elizaga ML, Vasan S, Marovich MA, Sato AH, Lawrence DN, Chaitman BR, Frey SE, Keefer MC; MVA Cardiac Safety Working Group. Prospective surveillance for cardiac adverse events in healthy adults receiving modified vaccinia Ankara vaccines: a systematic review. PLoS One. 2013;8(1):e54407. doi: 10.1371/journal.pone.0054407. Epub 2013 Jan 17. PMID 23349878
- [Derived] Walsh SR, Seaman MS, Grandpre LE, Charbonneau C, Yanosick KE, Metch B, Keefer MC, Dolin R, Baden LR. Impact of anti-orthopoxvirus neutralizing antibodies induced by a heterologous prime-boost HIV-1 vaccine on insert-specific immune responses. Vaccine. 2012 Dec 17;31(1):114-9. doi: 10.1016/j.vaccine.2012.10.093. Epub 2012 Nov 7. PMID 23142302
- [Derived] Keefer MC, Frey SE, Elizaga M, Metch B, De Rosa SC, Barroso PF, Tomaras G, Cardinali M, Goepfert P, Kalichman A, Philippon V, McElrath MJ, Jin X, Ferrari G, Defawe OD, Mazzara GP, Montefiori D, Pensiero M, Panicali DL, Corey L; NIAID HIV Vaccine Trials Network. A phase I trial of preventive HIV vaccination with heterologous poxviral-vectors containing matching HIV-1 inserts in healthy HIV-uninfected subjects. Vaccine. 2011 Feb 24;29(10):1948-58. doi: 10.1016/j.vaccine.2010.12.104. Epub 2011 Jan 7. PMID 21216311